CLINICAL TRIAL: NCT06274515
Title: A Multi Cohort Translational Research Study to Investigate Mechanisms of Resistance to Breast Cancer Therapies
Brief Title: A Study to Investigate Mechanisms of Resistance to Breast Cancer Therapies
Acronym: REMERGE
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WO44977
Record Dates: First submitted 2024-01-24; First posted 2024-02-23 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mechanisms of Acquired Resistance (Experimental): Participants with breast cancer who have a newly appearing or recurrent metastatic lesion while on anti-cancer therapy will be assigned to one of 3 cohorts.
  Interventions: Procedure: Tumor Tissue and Blood Draw
- Mechanisms of Primary Resistance (Experimental): Participants with breast cancer who have a progressing tumor lesion while on anti-cancer therapy will be assigned to one of 2 cohorts.
  Interventions: Procedure: Tumor Tissue and Blood Draw

INTERVENTIONS:
Procedure: Tumor Tissue and Blood Draw — Participants will have their blood drawn on the day a tissue sample is taken from a progressive tumor lesion.

SUMMARY:
This study will evaluate mechanisms of resistance to anti-breast cancer therapies in tumor and blood samples from participants with human epidermal growth factor receptor (HER2) positive, hormone receptor (HR) positive or triple negative breast cancer.

ELIGIBILITY:
General Inclusion Criteria:

* Willingness to undergo a procedure to obtain tumor tissue (e.g. biopsy) and blood draw
* Diagnosis of HER2+, HR+ (for cohort R1) or triple negative breast cancer (for cohort T1) as per local assessment
* Availability of an archival tumor tissue (most recent pre-treatment tumor tissue is preferred)
* Unequivocally growing tumor lesion (progressive lesion) that is accessible for resection, excision or core needle biopsy
* Discontinuation of prior anti-cancer treatment outlined below should not be longer than 4 weeks from participation in this study

Inclusion criteria for participants in the cohorts studying acquired resistance

* Participant had undergone regular monitoring for disease progression as per local practice (preferably every 3-6 months) while on most recent breast cancer therapy
* Accessible tumor lesion that newly appeared or a lesion that started to regrow while the participant was at least 6 months on therapy

Inclusion criteria for participants in the cohort studying primary resistance

* Accessible tumor lesion that continued to increase in size or a newly appearing lesion (as confirmed by routine tumor assessment) while treated for at least 4 weeks but less than 6 months on therapy

Exclusion Criteria:

* Any risks factors that increase the risk of complications associated with the procedure to obtain tumor tissue (e.g. bleeding disorders)
* Any serious medical condition or abnormality in clinical laboratory tests that precludes an individual's safe participation in and completion of the study
* Participant has started treatment with subsequent anti-cancer therapy
* Participants whose progressive tumor lesion that is targeted for biopsy/resection is in the bone
* Discontinuation of treatment was due to a reason other than disease progression

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2024-04-02 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in HER2 protein levels measured at the time of disease progression/recurrence (Cohorts H1 and H2) | At least 6 months
Changes from baseline in HER2 gene copy number measured at the time of disease progression/recurrence (Cohorts H1 and H2) | At least 6 months
Changes from baseline in estrogen receptor (ER) protein levels measured at the time of disease progression/recurrence (Cohorts H1 and H2) | At least 6 months
Changes from baseline in HER2 protein levels measured at the time of disease progression/recurrence (Cohort H3) | Less than 6 months
Changes from baseline in HER2 gene copy number measured at the time of disease progression/recurrence (Cohort H3) | Less than 6 months
Changes from baseline in ER protein levels measured at the time of disease progression/recurrence (Cohort H3) | Less than 6 months
Changes from baseline in genes related to CDK4/6 resistance (incl. cell cycle alterations and tyrosine kinase receptors, Cohort R1) | At least 6 months
Changes from baseline in genes related to endocrine resistance (incl. cell cycle alterations and tyrosine kinase receptors, Cohort R1) | At least 6 months
Changes from baseline in tumor immune microenvironment (PD-L1 and TILs, Cohort T1) | At least 6 months
Changes from baseline in immune phenotype (PD-L1 and TILs, Cohort T1) | At least 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (26):
- Belgium (3):
  - Institut Jules Bordet, Anderlecht
  - CHU de Liège (Sart Tilman), Liège
  - AZ Delta (Campus Rumbeke), Roeselare
- Denmark (2):
  - Aalborg Universitetshospital, Aalborg
  - Sjællands Universitetshospital, Næstved, Næstved
- Finland (2):
  - Helsinki University Central Hospital, Helsinki
  - Tampere University Hospital, Tampere
- Germany (4):
  - St. Elisabeth Krankenhaus Köln GmbH, Cologne
  - KEM/Evang. Kliniken Essen Mitte gGmbH, Essen
  - ViDia Christliche Kliniken Karlsruhe, Vincentius-Diakonissen-Kliniken gAG, Karlsruhe
  - Universitätsklinikum Mannheim, Mannheim
- Italy (7):
  - I.R.S.T Srl IRCCS, Meldola, Emilia-Romagna
  - Azienda Ospedaliero - Universitaria di Modena Policlinico, Modena, Emilia-Romagna
  - RCCS - Centro di Riferimento, Aviano (PN), Friuli Venezia Giulia
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Rome, Lazio
  - Ospedale San Raffaele S.r.l. - PPDS, Milan, Lombardy
  - Irccs Istituto Nazionale Dei Tumori (Int), Milan, Lombardy
  - Irccs Istituto Europeo Di Oncologia (IEO), Milan, Lombardy
- Oslo university hospital Radiumhospitalet, Oslo, Norway
- Spain (4):
  - Hospital Universitario 12 de Octubre, Madrid
  - HM Sanchinarro ? CIOCC, Madrid
  - Hospital Universitario Virgen del Rocio, Seville
  - Hospital Clínico Universitario de Valencia, Valencia
- United Kingdom (3):
  - Basingstoke and North Hampshire Hospital, Basingstoke
  - Imperial College Healthcare NHS Trust, London
  - Christie Hospital NHS Trust, Manchester

IPD SHARING:
Plan to Share IPD: No